CLINICAL TRIAL: NCT07378137
Title: A Preference Study Comparing the Components of Composite Endpoints for Healthcare Providers and Patients With CAD
Brief Title: Comparing the Components of Composite Endpoints for Healthcare Providers and Patients
Acronym: REC-CHARTENDS
Status: Recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Ling Tao, MD, PhD, Professor in Cardiology, Director of the Department of Cardiology, Xijing Hospital
Other Study IDs: REC-CHARTENDS
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease; Percutaneous Coronary Intervention
Keywords: coronary artery disease; composite endpoints
MeSH Terms: conditions — Coronary Artery Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects: Medical staff and patients with CAD
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — A questionnaire regarding the weights given by the patients with CAD and the medical staff for the individual components of the composite endpoint

SUMMARY:
Clinical trials often employ a composite primary endpoint to increase event rates and enhance trial efficiency. However, analytic approaches to composite endpoints typically assume that the individual components are of similar importance. In practice, a treatment often has different effects on each individual endpoint, leading to uncertainty in interpreting the results of a clinical trial employing a composite primary endpoint.

Some investigators have recommended using a weighted composite endpoint to address these concerns, in which individual components are valued relative to one another. However, data to inform the weighting of individual endpoints, using opinions from both medical staff and patients, remains controversial. Furthermore, prior efforts to weigh composite endpoints have assumed that patients, physicians, and clinical trialists would assign similar values to individual events. If patients value endpoints differently from trialists, this would suggest that efforts to develop weighted composite endpoints may also need to address patient preferences.

In the current study, we aim to record the weighing of both patients and medical staff towards a composite endpoint frequently used in cardiovascular clinical trials. To better understand the value of each endpoint for patients and medical staff, we quantified the relative severity of each endpoint when compared to death and assessed for rating differences between the two groups. Additionally, we investigated whether endpoint weights varied by the demographic and clinical characteristics of patients and medical staff.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute or chronic coronary syndrome who have undergone percutaneous coronary intervention;
2. Patients who can understand the purpose of this trial and are willing to participate in the preference questionnaire.
3. Healthcare providers who treat patients with coronary artery disease.

Exclusion Criteria:

1. Aged < 18 years;
2. Inability to understand the questionnaire or presence of cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthcare providers and patients with CAD
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Relative weight of myocardial infarction to death | Before discharge
Relative weight of stroke to death | Before discharge
Relative weight of cardiopulmonary resuscitation to death | Before discharge
Relative weight of procedural complications to death | Before discharge
Relative weight of major bleeding events to death | Before discharge
Relative weight of acute kidney injury to death | Before discharge
Relative weight of revascularization to death | Before discharge
Relative weight of rehospitalization to death | Before discharge

CONTACTS AND LOCATIONS:
Overall Officials: Ling Tao, M.D., Ph.D, Study Chair — Xijing Hospital; Chao Gao, M.D., Ph.D, Study Chair — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China